CLINICAL TRIAL: NCT03890133
Title: Exploration the Therapeutic Mechanism of Ba-Duan-Jin in the Treatment of Fibromyalgia by Improving Intestinal Microecology
Brief Title: Exploration the Mechanism of Ba-Duan-Jin Therapy in the Management of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, Deputy chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 81873294
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Ba-Duan-Jin; Gut microbiota; Mechanism
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ba-Duan-Jin group (Experimental): The participants will be guided by a research staff to do the Ba-Duan-Jin therapy for 50 minutes twice weekly for 12 weeks, in the outpatient section of the hospital; Pregabalin placebo treatment will be administered at bedtime once a day, starting at 150 mg for the first week, and increase to the dose of 300 mg from the second week. After one week, if 300 mg dose is tolerable, then maintain it for 10 additional weeks, if not, then go back to the 150 mg dose for 10 additional weeks.
  Interventions: Behavioral: Ba-Duan-Jin
- Pregabalin group (Active Comparator): Wellness education and muscle relaxation exercise program: This program will be held for 50 minutes twice weekly for twelve weeks, containing 10-minute wellness education, 10-minute doctor-patient discussion, and 30-minute guided muscle relaxation exercise.
  Active pregabalin capsules: As same usage as the placebo pregabalin capsules.
  Interventions: Drug: Pregabalin capsule
- Healthy control group (No Intervention)

INTERVENTIONS:
Behavioral: Ba-Duan-Jin — Ba-Duan-Jin is a common form of "self-healthcare" Qigong exercise that has been practiced by Chinese people for at least eight hundred years.It consists of eight sets of simple movements. By combining meditation with slow, graceful movements,deep breathing, and relaxation, Ba-Duan-Jin practitioners believe it has the ability to move vital energy (Qi) throughout the body. Ba-Duan-Jin is also considered to be a multicomponent intervention that integrates physical, psychosocial, emotional, spiritual, and behavioral elements. While the biological mechanisms remain unclear.
  Other Names: Baduanjin; Eight Brocades; Eight-Section Brocade
  Arms: Ba-Duan-Jin group
Drug: Pregabalin capsule — Pregabalin is one of the three medications (pregabalin, duloxetine, and milnacipran) that have been approved by the Food and Drug Administration (FDA) to treat fibromyalgia in US, and the only medicine that has been approved in China.
  Arms: Pregabalin group

SUMMARY:
Fibromyalgia (FM) is a chronic debilitating musculoskeletal pain syndrome. "Central sensitization" is an important mechanism of the disease. Recent studies have shown that "microbiome-gut-brain axis" imbalance may be one of the important mechanisms of "central sensitization". The purpose of this study was to investigate the therapeutic mechanism of Ba-Duan-Jin therapy in the treatment of fibromyalgia by improving intestinal microecology. The mechanism was evaluated by comparing the results of brain functional MRI (fMRI) and microbacterial analysis of the patients' stool pre and post treatment .

ELIGIBILITY:
Inclusion Criteria:

* meet the 1990 American College of Rheumatology (ACR) Research Classification Criteria for fibromyalgia and 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria;
* be between the ages of 18 to 70 years;
* not taking medication for FM for at least 4 weeks;
* no special eating habits.

Exclusion Criteria:

* had practiced Ba-Duan-Jin, Tai Chi, yoga or other forms of Qigong exercise within 12 months of their recruitment to the study;
* be less than 40mm of pain VAS score;
* had renal failure, severe depression or anxiety;
* had any poorly-controlled comorbid medical conditions, such as dementia, cancer, thyroid disease, inflammatory arthritis;
* pregnancy or planned pregnancy within the study period;
* patients residing more than 70 miles from the research site;
* patients with a history of head trauma;
* a smoker or drinker;
* contraindications for MRI,including metal implants, cardiac pacemaker,false tooth, surgical artery clips, metal tattoos or claustrophobia;
* patients with cerebral infarction or cerebral hemorrhage.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The change of the Visual Analogue Scale (VAS) for pain from baseline. | Baseline, week4, week8, week12, week24
  Pain VAS, range from 0 to 100 mm with higher score indicating more severe pain.

SECONDARY OUTCOMES:
Gut microbiota sequencing results by analyzing metagenomes of microbial genes | Baseline, week12
  Fecal samples are obtained from the experimental group and control group. After extracting DNA from fecal samoles, high-throughput Illumina sequencing, gene classification, abundance calculation, functional and metabolic annotation will be performed on the extracted DNA. The Bowtie2, BWA and Soap2 will be selected for the comparison software. The condition of comparison is to obtain the comparison results of 95% identity (and above).
Serum Brain Derived Neurotrophic Factor (BDNF) levels | Baseline, week12
  Serum BDNF levels were measured in healthy control group and FM patients
The change of the revised Fibromyalgia Impact Questionnaire (FIQR) from baseline. | Baseline, week 4, week 8, and week 12.
  A self-administered questionnaire with 10 subscales, measuring fibromyalgia symptoms and function domains. FIQR total score ranges from 0 to 100, with higher scores indicating more severe symptoms
Global Impression of Change (PGIC) questionnaire evaluated at week 12. | Week 12.
  A questionnaire determine any change in overall symptom status from the beginning of the study to its conclusion (score range, 1 [very much improved] to 7 [very much worse).
fMRI of the brain in patients with fibromyalgia | Baseline, week12
  To compare the changes in structure, connectivity and metabolic function of the brain in patients with fibromyalgia before and after treatment by fMRI.
Serum Tyrosine kinase B (TrkB) levels | Baseline, week12
  Serum TrkB levels were measured in healthy control group and FM patients

CONTACTS AND LOCATIONS:
Locations (1):
- GAMhospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiao J, Russell IJ, Wang W, Wang J, Zhao YY, Jiang Q. Ba-Duan-Jin alleviates pain and fibromyalgia-related symptoms in patients with fibromyalgia: results of a randomised controlled trial. Clin Exp Rheumatol. 2019 Nov-Dec;37(6):953-962. Epub 2019 Feb 15. PMID 30789154
- [Derived] Wu S, Jing B, Wang Y, Long M, Li Y, Li Z, Jiao J. Two Neuroanatomical Subtypes in Fibromyalgia Patients: Distinct Morphological Patterns and Treatment Outcomes. CNS Neurosci Ther. 2025 Jul;31(7):e70500. doi: 10.1111/cns.70500. PMID 40589353
- See also: Ba-Duan-Jin alleviates pain and fibromyalgia-related symptoms in patients with fibromyalgia: results of a randomised controlled trial. — https://pubmed.ncbi.nlm.nih.gov/30789154/